CLINICAL TRIAL: NCT00156663
Title: Toward Gender Aware VA Health Care: Development and Evaluation of an Intervention
Brief Title: Toward Gender Aware VA Healthcare: Development and Evaluation of an Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: GEN 20-057
Record Dates: First submitted 2005-08-25; First posted 2005-09-12 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Women's Health
Keywords: Women; Veterans; Delivery of Healthcare; Intervention Studies; United States Department of Veterans Affairs; Women's Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Caring for Women Veterans

INTERVENTIONS:
Behavioral: Caring for Women Veterans

SUMMARY:
The purpose of this study was to develop and evaluate an educational program intended to raise staff awareness about women veterans and their health care needs and preferences.

DETAILED DESCRIPTION:
OBJECTIVES:

The primary objective of this project was to develop and evaluate a computerized program that would enhance Veterans Health Administration (VHA) employees� awareness of women veterans and their health-care needs. The program was designed to challenge negative stereotypes about female patients (gender-role ideology), increase empathy toward female patients� needs (gender sensitivity), and enhance knowledge regarding women veterans and aspects of their VHA care (knowledge).

DESIGN/METHODS:

Phases I involved generating content for the computerized interactive program. Phase II involved creating the 30-minute program. The Phase III evaluation of the program involved a two-group pretest�posttest�follow-up equivalent control group design at two facilities with a third facility comparison group. At the first two facilities, employees who provide either direct or ancillary care to patients were randomly assigned to either the treatment or the control group. Participants in the treatment group completed the program entitled Caring for Women Veterans. Participants in the control group and those at the third site completed a 30-minute program entitled Managing Stress. The data from the third site were included to test for infusion of the treatment effect within same-site groups. Gender awareness was evaluated at three time points using the Gender Awareness Inventory-VA (GAI-VA). Participants completed the GAI-VA several weeks prior to completing the computerized program (Time 1, n =339), immediately after completing the program (Time 2, n = 249), and approximately one month after the program (Time 3, n = 167). Participants also completed a qualitative evaluation of the program at Time 2.

STATUS:

Complete.

ELIGIBILITY:
Inclusion Criteria:

Participants must be VHA employees who have direct or indirect contact with patients.

Exclusion Criteria:

Employees who have no contact with patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2004-05; Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Gender Awareness is measured during the pre-test, immediately after the educational program, and approximately four weeks after the subject participates in the educational program.

SECONDARY OUTCOMES:
Participants rate their enjoyment of the educational program and offer recommendations for the program as needed.

CONTACTS AND LOCATIONS:
Overall Officials: Dawne S Vogt, PhD BA, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA; Lynda A. King, PhD, Principal Investigator — VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA
Locations (2):
- United States (2):
  - Edith Nourse Rogers Memorial Veterans Hospital, Bedford, MA, Bedford, Massachusetts
  - VA Boston Healthcare System Jamaica Plain Campus, Jamaica Plain, MA, Boston, Massachusetts

REFERENCES:
- [Result] Vogt DS, Barry AA, King LA. Toward gender-aware health care: evaluation of an intervention to enhance care for female patients in the VA setting. J Health Psychol. 2008 Jul;13(5):624-38. doi: 10.1177/1359105308090934. PMID 18519436